CLINICAL TRIAL: NCT05339438
Title: Pre-operative Mapping of the Anterior Temporal Lobe Using Functional MRI Innovative Techniques in in Drug-resistant Epileptic Patients
Acronym: CARTA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Jacques JONAS, Principal Investigator, neurologist, Central Hospital, Nancy, France
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-A02968-33
Record Dates: First submitted 2022-04-06; First posted 2022-04-21 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Epilepsy, Temporal Lobe; Cognitive Decline
MeSH Terms: conditions — Epilepsy, Temporal Lobe; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epileptic patients (Experimental): Epileptic patients with anterior temporal lobe epilepsy
  Interventions: Radiation: functional MRI
- Healthy volunteers (Experimental): Healthy volunteers
  Interventions: Radiation: functional MRI

INTERVENTIONS:
Radiation: functional MRI — Functional MRI scanning (around 1h30 min): SMS + multi-band (with FPVS paradigms for both)

SUMMARY:
Anterior temporal epilepsy is the most frequent form of focal epilepsy (more than 50% of focal epilepsies). The epilepsy is drug-resistant when epileptic seizures persist despite antiepileptic treatment (25% of cases). In this case, it is possible to offer a surgical solution to the patient: an anterior temporal lobectomy. This surgery consists of removing the entire portion of the temporal lobe responsible for epilepsy (epileptogenic zone), that is to say a major part of the temporal pole, the hippocampus and the ventral anterior temporal lobe (vATL). The goal of the surgery is to lead to a disappearance of the seizures while preserving the functions of the patient. This is why a pre-surgical assessment is systematically carried out in order to locate the epileptic focus and to predict the risks of neurological and cognitive deficits. The vATL is of particular interest because it is a highly functional region, involved in naming, semantic processing and face recognition. A resection of this region by anterior lobectomy can therefore impact these functions and lead to cognitive deficits (for example, up to 65% decline in naming), which can be disabling in the lives of patients, even if they are free from seizures. One of the major challenges of epilepsy surgery is therefore to predict the postoperative neuropsychological outcome. The prediction of the neuropsychological outcome of the post-surgery patient is largely based on the mapping of functional regions preoperatively, carried out by functional MRI (fMRI), or by electrical stimulation carried out during intracerebral exploration by StereoElectroEncephalography (SEEG).

However, current techniques have drawbacks. Electrical stimulations are based on an invasive exploration (SEEG), are time-consuming and sometimes difficult to interpret. The fMRI sequences used in clinical routine do not make it possible to visualize the entire vATL region because of artifacts related to the auditory canal. Thus, the signal is strongly diminished in this region, rendering a large area of the vATL invisible. This results in insufficient visualization of activated vATL regions when performing tasks such as naming, semantic processing, and face recognition. Important functional regions can therefore be removed during surgery and negatively impact the patient's neuropsychological outcome.

In the CARTA study, original methods are associated in order to increase the signal-to-noise ratio in vATL. On the one hand, the Multi-Band sequence, an innovative fMRI sequence, will be used. On the other hand, a particular method of presentation of visual stimuli will be used, called fast periodic visual stimulation (FPVS: Fast Periodic Visual Stimulation), during which the stimuli are presented periodically (fixed frequency). Individually, these methods improve vATL (signal enhancement) exploration. The investigators assume that the combination of the two methods may have a potentiating effect, compared to the standard SMS (Simultaneous Multi-Slice) sequence. fMRI exploration will not influence the surgical management of the patient included in the study because it is the beginning of the development of this technique, but could be used, in the longer term, to guide the surgeries of epileptic patients.

Thus, the goal of this study is to precisely map the vATL, using innovative methods in fMRI. This mapping will make it possible to study the cerebral functions of the vATL involved in naming, semantic processing and face recognition, and ultimately improve the postoperative neuropsychological prognosis of epileptic patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult person,
* Person affiliated to a social security scheme or beneficiary of such a scheme,
* Person having received complete information on the organization of the Clinical Investigation and having signed informed consent,
* Person having carried out a preliminary clinical examination adapted to the Clinical Investigation,
* For patients: Person with drug-resistant structural focal epilepsy of the anterior temporal lobe (right or left), candidate for epilepsy surgery (anterior temporal lobectomy),
* For healthy volunteers: Person with no known pathology in the anterior temporal lobe (particularly epilepsy).

Exclusion Criteria:

* Contraindication to MRI including claustrophobia,
* Uncorrected visual disturbances,
* Person unable to give consent,
* Lack of mastery of the French language or ability to understand instructions,
* Person referred to in Articles 64, 65 and 66 of European Regulation 2017/745: Person of full age unable to consent alone to participate in the Clinical Investigation; Minor; Pregnant or breastfeeding woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-10 (Actual); Primary Completion 2027-06-09 (Estimated); Study Completion 2027-06-09 (Estimated)

PRIMARY OUTCOMES:
Functional Anterior Temporal Lobe activity | 3 years
  Blood Oxygen Level Dependent (BOLD) measures for each task (naming, semantic processing, and face recognition)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Régional Universitaire de Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Visser M, Lambon Ralph MA. Differential contributions of bilateral ventral anterior temporal lobe and left anterior superior temporal gyrus to semantic processes. J Cogn Neurosci. 2011 Oct;23(10):3121-31. doi: 10.1162/jocn_a_00007. Epub 2011 Mar 10. PMID 21391767
- [Result] Jonas J, Jacques C, Liu-Shuang J, Brissart H, Colnat-Coulbois S, Maillard L, Rossion B. A face-selective ventral occipito-temporal map of the human brain with intracerebral potentials. Proc Natl Acad Sci U S A. 2016 Jul 12;113(28):E4088-97. doi: 10.1073/pnas.1522033113. Epub 2016 Jun 27. PMID 27354526
- [Result] Jonas J, Rossion B, Brissart H, Frismand S, Jacques C, Hossu G, Colnat-Coulbois S, Vespignani H, Vignal JP, Maillard L. Beyond the core face-processing network: Intracerebral stimulation of a face-selective area in the right anterior fusiform gyrus elicits transient prosopagnosia. Cortex. 2015 Nov;72:140-155. doi: 10.1016/j.cortex.2015.05.026. Epub 2015 Jun 4. PMID 26143305
- [Result] Puckett AM, Bollmann S, Poser BA, Palmer J, Barth M, Cunnington R. Using multi-echo simultaneous multi-slice (SMS) EPI to improve functional MRI of the subcortical nuclei of the basal ganglia at ultra-high field (7T). Neuroimage. 2018 May 15;172:886-895. doi: 10.1016/j.neuroimage.2017.12.005. Epub 2017 Dec 5. PMID 29208571
- [Result] Gao X, Gentile F, Rossion B. Fast periodic stimulation (FPS): a highly effective approach in fMRI brain mapping. Brain Struct Funct. 2018 Jun;223(5):2433-2454. doi: 10.1007/s00429-018-1630-4. Epub 2018 Mar 3. PMID 29502144